CLINICAL TRIAL: NCT06863220
Title: Intravesical Ozone Therapy for Interstitial Cystitis/Bladder Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, urologist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 340434043404
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial Cystitis; bladder pain syndrome; ozone therapy; intravesical ozone
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ozone Therapy Group (Experimental): Patients received 50 mL ozonated saline (20-40 µg/mL) intravesically twice weekly for 3 weeks.
  Interventions: Other: Intravesical Ozone Therapy
- Placebo Group (Placebo Comparator): Patients received 50 mL normal saline intravesically twice weekly for 3 weeks.
  Interventions: Other: Placebo (Normal Saline)
- Control Group (Other): Patients continued standard care (e.g., oral pentosan polysulfate) without intravesical intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intravesical Ozone Therapy — Patients received 50 mL ozonated saline (20-40 µg/mL) intravesically twice weekly for 3 weeks.
  Arms: Ozone Therapy Group
Other: Placebo (Normal Saline) — Patients received 50 mL normal saline intravesically twice weekly for 3 weeks.
  Arms: Placebo Group
Other: Control — Patients continued standard care (e.g., oral pentosan polysulfate) without intravesical intervention.
  Arms: Control Group

SUMMARY:
This randomized, double-blind, placebo-controlled trial evaluated the efficacy and safety of intravesical ozone therapy in 60 patients with interstitial cystitis (IC). Participants were assigned to ozone therapy, placebo, or standard care groups for 3 weeks, with follow-up at 6 weeks. The primary outcome was the change in O'Leary-Sant ICSI score. Secondary outcomes included VAS pain score, SF-36 physical health, and urinary frequency.

DETAILED DESCRIPTION:
Patients received either 50 mL ozonated saline (20-40 µg/mL), normal saline (placebo), or continued standard care twice weekly for 3 weeks. Assessments were conducted at baseline, week 3, and week 6. The study aimed to determine if ozone therapy reduces interstitial cystitis symptoms compared to placebo and standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Histopathologically or clinically confirmed IC (per AUA guidelines)
* Symptoms for at least 6 months
* Willing to provide informed consent

Exclusion Criteria:

* Active urinary tract infection
* Bladder malignancy
* Pregnancy or breastfeeding
* Known ozone allergy
* Intravesical therapy within 3 months
* G6PD deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in O'Leary-Sant ICSI Score | Baseline to Week 3
  Reduction in symptom severity measured by the O'Leary-Sant Interstitial Cystitis Symptom Index (range 0-19).

SECONDARY OUTCOMES:
VAS pain score | baseline to week 3
  Reduction in pelvic pain measured by Visual Analog Scale (range 0-10).
Change in Daily Urinary Frequency | baseline to week 3
  Reduction in average daily voiding frequency via 3-day voiding diary.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to privacy concerns and the absence of a data-sharing agreement.

REFERENCES:
- [Background] Pires MV, de Lima CJ, Carvalho HC, Moreira LH, Fernandes AB. Effectiveness of intravesical ozone in interstitial cystitis by the O'Leary-Sant symptom index. Int Urogynecol J. 2023 Jul;34(7):1437-1446. doi: 10.1007/s00192-022-05383-3. Epub 2022 Oct 15. PMID 36242631